CLINICAL TRIAL: NCT06995443
Title: Breast Cancer and Chemobrain : Effects of Photobiomodulation on the Improvement of Perceived Cognitive Impairment - REGAIN
Brief Title: Breast Cancer and Chemobrain : Effects of Photobiomodulation on the Improvement of Perceived Cognitive Impairment
Acronym: REGAIN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier de Valenciennes (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2024-02-02
Record Dates: First submitted 2025-02-26; First posted 2025-05-29 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Oncology; Support Care; Cognitive Disorders
Keywords: Cognitive disorders; Photobiomodulation; Breast cancer; oncology
MeSH Terms: conditions — Neoplasms; Cognitive Dysfunction; Breast Neoplasms | interventions — Low-Level Light Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care with photobiomodulation sessions (Experimental): Photobiomodulation : 1 session per week during 12 weeks Visit 1 to Visit 4 : Photobiomodulation (NOVOTHOR) + cortical stimulation (VEILIGHT) Visit 5 to 12 : Cortical stimulation Visit 13 (V12 + 7 days +/- 3 days) : FACT-COG / anxiety measure / depression measure / Likert scale / satisfaction Visit 6 months (V1 + 6M +/- 2 weeks) : questionnary FACT-COG
  Interventions: Other: Photobiomodulation
- Usual care (No Intervention)

INTERVENTIONS:
Other: Photobiomodulation — 12 sessions of photobiomodulation (1 per week) Visit 1 to 4 : photobiomodulation (NOVOTHOR) + cortical stimulation (VEILIGHT) Visit 5 to 12 : cortical stimulation (VEILIGHT)
  Arms: Usual care with photobiomodulation sessions

SUMMARY:
Breast cancer is one of the most common cancers in metropolitan France, with over 60,000 new cases in 2023. Mostly a female cancer, it can affect a young population, with around 20% of breast cancers occurring in women under 50. Treatment is mainly based on surgery, chemotherapy, radiotherapy, targeted therapies and hormone therapy. Although chemotherapy is not systematically used, it remains a frequent treatment option. While chemotherapy makes a major contribution to curing cancer, it is also a source of potentially disabling side effects for survivors.

Chemotherapy can interfere with the normal functioning of the central nervous system, leading to cognitive impairment. The number of people potentially affected by chemobrain is estimated at several tens of millions worldwide. There is no recommended treatment for people with chemobrain. Several avenues have been explored, with very limited results. Photobiomodulation (PBM) is a non-medicinal treatment technique that combines all the biological, athermic and non-cytotoxic effects of tissue exposure to non-ionizing sources of red and infrared light. Several studies have demonstrated the beneficial effects of cortical stimulation by photobiomodulation on memory (increased angiogenesis, increased oxygenation of brain tissue via vasodilatation, and increased mitochondrial ATP production). These positive biological effects are likely to ameliorate the undesirable effects of chemotherapy, and consequently the post-chemotherapy cognitive disorders that ensue.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 and over
* Having completed chemotherapy (intravenous) for breast cancer (any stage) less than 12 months prior to inclusion
* Having a perceived cognitive complaint that appeared during or after (< 3 months) chemotherapy treatments (no restriction on the care protocol used) and confirmed by a FACT-Cog score compatible with a subjective cognitive disorder (score < 117 for patients aged 18 to 49; score < 113 for patients aged 50 to 69; score <105 for patients aged 70 and over)
* Patient eligible for photobiomodulation sessions
* Patient with sufficient command of the French language to complete the study questionnaries
* Patient having given written consent to participate in the trial
* Socially insured patient
* Patient willing to comply with all study procedures and duration

Exclusion Criteria:

* Known cognitive disorders prior to chemotherapy treatment
* Patients with psychiatric or psychobehavioral disorders incompatible with photobiomodulation sessions
* Patients who, in the 12 months prior to inclusion or at the time of inclusion, have already received photobiomodulation treatment involving "whole body" therapy (photobiomodulation in a phototherapy booth).
* Patient having previously received photobiomodulation with cortical stimulation (panel or helmet) with no time limit.
* Patient taking or having received capecitabine
* Patients taking part in a protocol involving a drug likely to affect cognitive performance (on the investigator's advice).
* Patients suffering from claustrophobia
* Patient unable to read and/or unable to complete a questionnaire, in the opinion of the investigator

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Women aged 18 years and over
Enrollment: 200 (Estimated)
Dates: Start 2025-06-13 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
To compare, among women aged 18 and over who had undergone chemotherapy for breast cancer and had subjective cognitive impairment post-chemotherapy, the rate of those showing improvement in cognitive impairment with or without photobiomodulation (cortica | From enrollment to the end of follow-up visit at 13 weeks (V13 = V12 + 7d +/- 3d)
  Patients with an evolution subjective cognitive performance between the FACT-Cog performed at inclusion and that at the end of follow-up (S13)

SECONDARY OUTCOMES:
Compare the rate of patients considered anxious in each group at inclusion (T0) and at the end of the follow-up period (S13) | From enrollment to the end of follow-up visit at 13 weeks (V13 = V12 + 7d +/- 3d)
  For patients aged 18 to 65: HAD anxiety score (first 7 questions, score variable from 0 to 21).
  For patients > 65 years: GAI FC SF score (5 questions, score variable from 0 to 5).
  The cut-off will be 8 for the HAH anxiety score and 3 for the GAI FC SF
To compare the rate of patients considered depressed in each group at inclusion (T0) and at the end of the follow-up period (S13) | From enrollment to the end of follow-up visit at 13 weeks (V13 = V12 + 7d +/- 3d)
  For patients aged 18 to 65: HAD depression score (last 7 questions, score variable from 0 to 21).
  For patients > 65 years: mini-GDS score (5 questions, score variable from 0 to 5).
  The cut-off will be 8 for the HAD anxiety score and 1 for the GAI FC SF
Compare perceived sleep quality in each group at inclusion (T0) and at the end of the follow-up period (13) | From enrollment to the end of follow-up visit at 13 weeks (V13 = V12 + 7d +/- 3d)
  Perceived sleep on a Likert scale by answering the question "How would you rate the quality of your sleep: very good, good, bad, very bad"
Compare perceived health in each group at inclusion (T0) and at the end of the follow-up period (S13) | From enrollment to the end of follow-up visit at 13 weeks (V13 = V12 + 7d +/- 3d)
  Perceived health on a Likert scale by answering the question "How would you rate your health: very good, good, bad, very bad"
Describe in the experimental group only the evolution of the FACT-Cog score at the end of photobiomodulation treatment (S13) and at 6 months | From follow-up visit at 13 weeks and 6 months after the first session of photobiomodulation (V1 + 6M +/-2W)
  Overall FACT-Cog score at S13 and 6-month follow-up
Evaluate the level of satisfaction of patients in the intervention group regarding the course of PBM sessions | At the follow-up visit V13 (=V12 + 7d +/- 3d)
  Level of satisfaction with various aspects of the sessions on a Likert scale by answering the following questions:
  - Concerning the frequency of photobiomodulation sessions: "How would you rate your satisfaction on a scale from 0 (not satisfied at all) to 10 (completely satisfied)?
  - Concerning duration: "How would you rate your satisfaction on a scale from 0 (not satisfied at all) to 10 (completely satisfied)?
  - Concerning the organization of photobiomodulation sessions: "How would you rate your satisfaction on a scale from 0 (not satisfied at all) to 10 (completely satisfied)?

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier de Valenciennes, Valenciennes, France